CLINICAL TRIAL: NCT00673244
Title: Protocol to Assess the Severity of Acute Kidney Injury
Acronym: AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB# 010835
Record Dates: First submitted 2008-04-15; First posted 2008-05-07 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Failure
Keywords: Renal Replacement Therapy; Dialysis
MeSH Terms: conditions — Acute Kidney Injury | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — One dose: 1 mg/kg (iv)if the patient is furosemide naive or 1.5 mg/kg (iv) if patient is not furosemide naive.
  Other Names: Lasix

SUMMARY:
The principal objective is to safely determine if we can identify the severity of Acute Kidney Injury (AKI) early in the course of the disease. Once enrolled, we will draw blood and urine for relevant biomarkers. Our goal is to validate if any of these biomarkers can predict the course of AKI (recovery v. RRT v. death)

DETAILED DESCRIPTION:
AKI is a very common disease in the intensive care unit. However, despite advances in supportive care, patients with AKI carry a high mortality rate (50% to 70%). The established AKI affects nearly 5 percent of hospitalized persons and as many as 15 percent of critically ill patients. Currently, there are no FDA approved therapeutic agents for the treatment of AKI.

Retrospective studies suggest that the early initiation of renal replacement therapy (RRT) improves outcome. Many clinicians tend to take a "wait and see" approach because they do not want to dialyze a patient who is destined to recover renal function without the need for RRT. Therefore, it is vitally important to know early in the course which patients with AKI are likely to progress to RRT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Increase in serum creatinine of 0.3 mg/dl within 48 hours or an increase of greater or equal to 150 to 200% from baseline or sustained oliguria(mean urine output of <0.5 cc/kg/hr for 6 hours within 48 hours)
* Written informed consent
* Patients who already have a indwelling bladder catheter

Exclusion Criteria:

* Voluntary refusal or missing written consent of the patient or the designated legal representative
* Patients with advanced Chronic Kidney Disease - as defined by a baseline GFR of < 30 ml/min as calculated by the MDRD equation
* Patients with renal transplantation
* Pregnancy
* Patients with an allergy or sensitivity to loop diuretics
* Patients with a clinical syndrome consistent with pre-renal AKI

  * Defined by fractional excretion of Na of < 1% AND no evidence of the urinary casts, or
  * Patients that are under-resuscitated as deemed by treating clinical team or
  * Patients who are actively bleeding
* Patients with a clinical syndrome of post-renal AKI

  * Any radiological study that shows hydro-ureter, or
  * Clinical scenario wherein the obstruction is considered a likely possibility of the cause of AKI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakmir S Chawla, MD, Principal Investigator — George Washigton University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Hou SH, Bushinsky DA, Wish JB, Cohen JJ, Harrington JT. Hospital-acquired renal insufficiency: a prospective study. Am J Med. 1983 Feb;74(2):243-8. doi: 10.1016/0002-9343(83)90618-6. PMID 6824004
- [Background] Liu KD, Himmelfarb J, Paganini E, Ikizler TA, Soroko SH, Mehta RL, Chertow GM. Timing of initiation of dialysis in critically ill patients with acute kidney injury. Clin J Am Soc Nephrol. 2006 Sep;1(5):915-9. doi: 10.2215/CJN.01430406. Epub 2006 Jul 6. PMID 17699307
- [Background] PARSONS FM, HOBSON SM, BLAGG CR, McCRACKEN BH. Optimum time for dialysis in acute reversible renal failure. Description and value of an improved dialyser with large surface area. Lancet. 1961 Jan 21;1(7169):129-34. doi: 10.1016/s0140-6736(61)91309-5. No abstract available. PMID 13733013
- [Background] Fischer RP, Griffen WO Jr, Reiser M, Clark DS. Early dialysis in the treatment of acute renal failure. Surg Gynecol Obstet. 1966 Nov;123(5):1019-23. No abstract available. PMID 5926520
- [Background] Kleinknecht D, Jungers P, Chanard J, Barbanel C, Ganeval D. Uremic and non-uremic complications in acute renal failure: Evaluation of early and frequent dialysis on prognosis. Kidney Int. 1972 Mar;1(3):190-6. doi: 10.1038/ki.1972.26. No abstract available. PMID 4545907
- [Background] Conger JD. A controlled evaluation of prophylactic dialysis in post-traumatic acute renal failure. J Trauma. 1975 Dec;15(12):1056-63. doi: 10.1097/00005373-197512000-00003. No abstract available. PMID 1202238
- [Background] Gettings LG, Reynolds HN, Scalea T. Outcome in post-traumatic acute renal failure when continuous renal replacement therapy is applied early vs. late. Intensive Care Med. 1999 Aug;25(8):805-13. doi: 10.1007/s001340050956. PMID 10447537
- [Background] Demirkilic U, Kuralay E, Yenicesu M, Caglar K, Oz BS, Cingoz F, Gunay C, Yildirim V, Ceylan S, Arslan M, Vural A, Tatar H. Timing of replacement therapy for acute renal failure after cardiac surgery. J Card Surg. 2004 Jan-Feb;19(1):17-20. doi: 10.1111/j.0886-0440.2004.04004.x. PMID 15108784
- [Background] Elahi MM, Lim MY, Joseph RN, Dhannapuneni RR, Spyt TJ. Early hemofiltration improves survival in post-cardiotomy patients with acute renal failure. Eur J Cardiothorac Surg. 2004 Nov;26(5):1027-31. doi: 10.1016/j.ejcts.2004.07.039. PMID 15519198
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219

RESULTS

PARTICIPANT FLOW:
Groups:
- Did Not Progress to AKIN Stage III: Did not meet the following criteria within 14 days of furosemide stress test (FST): Need for RRT, increase in serum creatinine of 300% over baseline, urine output of 0.3 cc/kg/hour × 24 hours
- Progressed to AKIN Stage III: Meet the following criteria within 14 days of Furosemide stress test (FST): need for RRT, increase in serum creatinine of 300% over baseline, urine output of 0.3 cc/kg/hour × 24 hours
Period: Overall Study
Arm/Group | Did Not Progress to AKIN Stage III | Progressed to AKIN Stage III
Started | 52 | 25
Completed | 52 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Did Not Progress to AKIN Stage III: Subject did not require RRT, increase in serum creatinine of 300% over baseline, urine output of 0.3 cc/kg/hour × 24 hours within 14 days of FST.
- Progressed to AKIN Stage III: Subject required RRT, increase in serum creatinine of 300% over baseline, urine output of 0.3 cc/kg/hour × 24 hours within 14 days of FST.
- Total: Total of all reporting groups
Arm/Group | Did Not Progress to AKIN Stage III | Progressed to AKIN Stage III | Total
Number analyzed (Participants) | 52 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (2.2) | 68.2 (1.9) | 65.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 11 | 44
  Male | 19 | 14 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 29 | 15 | 44
  Caucasian | 15 | 8 | 23
  Hispanic | 8 | 2 | 10
Chronic kidney disease [Count of Participants; unit: Participants] | 17 | 7 | 24
Hypertension [Count of Participants; unit: Participants] | 41 | 19 | 60
Congestive heart failure [Count of Participants; unit: Participants] | 15 | 10 | 25
Diabetes [Count of Participants; unit: Participants] | 22 | 13 | 35
NSAIDS [Count of Participants; unit: Participants] | 6 | 2 | 8
Aminoglycosides [Count of Participants; unit: Participants] | 0 | 1 | 1
Amphotericin [Count of Participants; unit: Participants] | 2 | 0 | 2
Contrast [Count of Participants; unit: Participants] | 15 | 6 | 21
Post-cardiac surgery [Count of Participants; unit: Participants] | 6 | 3 | 9
Sepsis [Count of Participants; unit: Participants] | 12 | 3 | 15
Baseline eGFR [Mean (Standard Deviation); unit: ml/minute/1.73m2] | 60.6 (8.8) | 73.3 (4.2) | 68.6 (4.1)
Baseline UFR [Mean (Standard Deviation); unit: ml/hr] | 95.7 (16.3) | 29.7 (4.2) | 74.6 (11.6)
Furosemide-naïve [Count of Participants; unit: Participants] | 23 | 6 | 29
Urinary Sediment Cast Scoring Index for Acute Kidney Injury [Mean (Standard Deviation); unit: Scores on a scale] — Urinary Sediment Cast Scoring Index is a biomarker for acute tubular necrosis which is the most common causes of acute kidney injury in hospitalized patients. Scores range from 1 to 4 with 1 being the best (no acute tubular necrosis) and 4 being the worst (severe acute tubular necrosis).
  1. No granular/epithelial cell casts
  2. Rare
  3. Moderate
  4. Sheets of muddy brown casts Chawla LS, Dommu A, Berger A, Shih S, Patel SS: Urinary sediment cast scoring index for acute kidney injury: a pilot study. Nephron Clin Pract 2008, 110:c145-150.
  Scores on a scale | 2.1 (0.16) | 2.7 (0.23) | 2.3 (0.13)
FeNa above 1% [Count of Participants; unit: Participants] | 10 | 4 | 14
Cardiovascular Sequential Organ Failure Assessment [Mean (Standard Deviation); unit: Scores on a scale] — This is sub-score of the sequential organ failure assessment score. Scores range from 0 (best) to 4 (worst).
  0: MAP ≥ 70 mmHg, no vasopressors
  1. MAP < 70 mmHg, no vasopressors
  2. dopamine ≤ 5 μg/kg/min or dobutamine (any dose)
  3. dopamine > 5 μg/kg/min OR epinephrine ≤ 0.1 μg/kg/min OR norepinephrine ≤ 0.1 μg/kg/mi
  4. dopamine > 15 μg/kg/min OR epinephrine > 0.1 μg/kg/min OR norepinephrine > 0.1 μg/kg/min
  Scores on a scale | 1.05 (0.2) | 1.5 (0.4) | 1.16 (0.3)
APACHE II score [Mean (Standard Deviation); unit: Scores of a scale] — APACHE II ("Acute Physiology And Chronic Health Evaluation II") is a severity-of-disease classification system. The score is an integer from 0 to 71 is computed based on 12 routine physiological measurements. Higher scores correspond to more severe disease and a higher risk of death.
  Scores of a scale | 16.5 (1.2) | 21.6 (2.5) | 17.8 (1.11)
AKIN stage at enrollment [Count of Participants; unit: Participants] — The AKIN classification system uses creatinine and urine output to classify the severity of acute kidney injury. The stages range from 0 to 3. 0 means no acute kidney injury. 3 means most severe acute kidney injury.
  1. Creatinine 1.5 - 2.0x from baseline or creatinine increased by at least 26.4μmol/L or u/o < 0.5ml/kg/hr × 6 hours
  2. Creatinine 2.0-3.0x from baseline or u/o < 0.5ml/kg/hr × 12 hrs 3 Creatinine > 3.0x from baseline or creatinine over 354 μmol/L with an acute increase by at least 44 μmol/L or u/o < 0.3ml/kg/hr × 24 hrs or anuria for 12 hours or initiation of RRT
  Participants
    AKIN I | 34 | 7 | 41
    AKIN II | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Urine Volume
Description: Urine output measured in ml/hr for first 6 hours after furosemide administration
Time Frame: Time from furosemide administration to 6 hours after furosemide administration
Measure: Mean (Standard Error); unit: ml
Groups:
- Progressed to AKIN Stage III: Need for RRT, increase in serum creatinine of 300% over baseline, urine output of 0.3 cc/kg/hour × 24 hours within 14 days of furosemide stress test.
- Did Not Progress to AKIN Stage-III: Did not need RRT, have increase in serum creatinine of 300% over baseline, or have urine output of 0.3 cc/kg/hour × 24 hours within 14 days of furosemide stress test.
Arm/Group | Progressed to AKIN Stage III | Did Not Progress to AKIN Stage-III
Number analyzed (Participants) | 25 | 52
ml
  Urine Volume - Hour 1 | 89 (33) | 329 (46)
  Urine Volume - Hour 2 | 96 (46.6) | 392 (42.2)
  Urine Volume - Hour 3 | 109 (35.4) | 311 (31.7)
  Urine Volume - Hour 4 | 88 (23.4) | 265 (31.1)
  Urine Volume - Hour 5 | 83 (23.7) | 219 (22.8)
  Urine Volume - Hour 6 | 75 (17.4) | 194 (22.3)

ADVERSE EVENTS:
Time Frame: 14 days after furosemide stress test or until hospital discharge
Groups:
- Progressed to AKIN III: RRT, increase in serum creatinine of 300% over baseline, urine output of 0.3 cc/kg/hour × 24 hours within 14 days of furosemide stress test
- Did Not Progress to AKIN III: No RRT, increase in serum creatinine of 300% over baseline, urine output of 0.3 cc/kg/hour × 24 hours within 14 days of furosemide stress test
Arm/Group | Progressed to AKIN III | Did Not Progress to AKIN III
All-Cause Mortality (participants affected / at risk) | 9/25 | 7/52
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/52
Other Adverse Events (participants affected / at risk) | 0/25 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No